CLINICAL TRIAL: NCT02997475
Title: Neural Bases of Multiple Forms of Self-regulatory Control in Bulimia Nervosa
Acronym: SRBN
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); The Hilda & Preston Davis Foundation (Other)
Responsible Party: Principal Investigator, Walter Kaye, Principal Investigator, University of California, San Diego
Other Study IDs: 151514; F32MH108311 (NIH)
Record Dates: First submitted 2016-10-25; First posted 2016-12-20 (Estimated); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia Nervosa; Bulimia; fMRI; Emotion Regulation; Response Inhibition
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Women with Bulimia Nervosa
- Women Healthy Controls

SUMMARY:
The purpose of this study is to investigate areas of the brain responsible for self-regulation in adult women who have never had an eating disorder with women who have bulimia nervosa. More specifically, investigators are interested in changes in brain activation (e.g., changes in blood flow and oxygen use) when inhibiting responses and regulating emotions. Data collection will rely on a technology called functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
General Inclusion Criteria:

* Female
* Right-handed
* Between the ages of 18 and 35 years

  *For Women with Bulimia Nervosa:
* Binge eating (i.e., eating a large amount of food while experiencing a sense of loss of control)
* Purging via self-induced vomiting (other methods may also be endorsed)

General Exclusion Criteria:

* Current significant medical illness or condition (e.g., diabetes, thyroid disease)
* Pregnancy, planned pregnancy, or lactation during the study period
* Non-removable metallic objects in the body

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women (ages 18-35 years) with bulimia nervosa, and age- and BMI-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2016-06; Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Self-Regulatory Control | Day 2 (fMRI Scan)
  Functional Magnetic Resonance Imaging will be used to assess brain activation associated with motor inhibitory control and affect regulation in women with bulimia nervosa (BN)

SECONDARY OUTCOMES:
Goal-Directed Action Control | Day 1
  An computerized instrumental learning task will be used to assess performance of women with and without bulimia nervosa.
Eating Disorder Relevance | Day 0
  The Eating Disorder Examination (EDE) will be conducted to assess relative associations of motor, affective, and goal-directed action control with bulimia nervosa severity.

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Berner, Ph.D., Study Director — University of California, San Diego
Locations (1):
- UCSD Eating Disorders Center for Treatment and Research, San Diego, California, United States